CLINICAL TRIAL: NCT05014555
Title: Sustained Humoral and Cell-Mediated Immunogenicity of COVID-19 Vaccines in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GI Alliance (Other)
Collaborators: Janssen, LP (Industry); University of Wisconsin, Madison (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CNTO1275IBD4005
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A Non-biologic Group: Participants on treatment regimen of mesalamine monotherapy or thiopurine monotherapy, or corticosteroids.
  Interventions: Biological: COVID-19 Vaccine
- Group B Anti-TNF Group: Participants on treatment regimen of maintenance montherapy of infliximab (at least 8 every 8 weeks), golilumamb (at least monthly), adalimumab (at least every 2 weeks), or certolizumab (at least monthly), or combination therapy of anti-TNF therapy as described above along with either 15mg of methotrexate or azathiprine at least 1.0mg/kg or 6MP 0.5mg/kg.
  Interventions: Biological: COVID-19 Vaccine
- Group C Ustekinumab Group: Participants on treatment regimen of ustekinumab monotherapy or combination therapy with methotrexate or azathioprine.
  Interventions: Biological: COVID-19 Vaccine
- Group D Vedolizumab Group: Participants on vedolizumab monotherapy or combination therapy with methotrexate or azathioprine.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Three-dose mRNA COVID-19 vaccine per standard of care

SUMMARY:
The aim of this study is to determine the impact of systemic immunosuppression on sustained antibody COVID-19 concentrations in patients with IBD who received a COVID-19 vaccine.

ELIGIBILITY:
A patient will be eligible for inclusion in this study if he or she meets all the following criteria:

* Patient is between the ages of 18-85 years, inclusive
* Patient has a history of ulcerative colitis (UC), or Crohn's disease diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria
* On one of the following treatment regimens for at least three months at the time of immunization and continued same therapy at the time of recruitment. Should be on stable doses defined as: Group A should have taken a dose of medication within the past week; Group B infliximab within the previous 8 weeks, golimumab within the previous 4 weeks, adalimumab within the previous 2 weeks, or certolizumab within the previous 4 weeks; Those on combination therapy in group B will have taken azathioprine or methotrexate within the past week. Group C ustekinumab at least within the previous 4 weeks. Those on combination therapy in group C will have taken azathioprine or methotrexate within the past week; Group D vedolizumab at least within the previous 4 weeks. Those on combination therapy in group D will have taken azathioprine or methotrexate within the past week

  * Group A non-biologic group: mesalamine monotherapy or thiopurine monotherapy
  * Group B: Anti-TNF Therapy Group: on maintenance therapy infliximab (at least 5mg/kg every 8 weeks), golimumab (at least monthly), adalimumab (at least every 2 weeks), or certolizumab (at least monthly Combination Therapy Anti- TNF Combination Therapy Group: on anti-TNF therapy as described above along with either 15mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg at least 40% of the group; Approximately 40-50% of the group will be combination therapy
  * Group C: Ustekinumab on either ustekinumab monotherapy or combination therapy with methotrexate or azathioprine
  * Group D: Vedolizumab Therapy Group: Vedolizumab Therapy: on either vedolizumab monotherapy or combination therapy with methotrexate or azathioprine
* Patient received at least two doses of mRNA COVID-19 vaccine per standard of care

A patient will not be eligible for inclusion in this study if he or she meets all the following criteria:

* Patient cannot or will not provide written informed consent
* Unable to provide appropriate informed consent due to being illiterate or impairment in decision-making capacity
* Received a COVID-19 booster within the previous 28 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease patients, Gastroenterology practice
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-05 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the immunogenicity of the COVID-19 vaccines by measuring geometric mean titers (GMT) of SARS-CoV-2 antibody concentrations, and quantitative assays to evaluate RBD-binding IgG levels | 6 and 12 months after third dose of the COVID-19 vaccine, with primary outcome being sustained antibody concentrations at 12 months
  Evaluation of the immunogenicity of the COVID-19 vaccines prior to patients receiving a COVID-19 booster during the Fall 2023 through Spring 2024 and at approximately six months after the Fall2023/Spring 2024 COVID-19 booster. Quantitative assays will be used to evaluate RBD-binding IgG levels.

SECONDARY OUTCOMES:
Sustained cell-mediated immunity against Covid-spike proteins will be evaluated using IFN-ϒ ELISpot, which detects both CD4 and CD8 T cell effectors. | during the Fall 2023 through Spring 2024 and at approximately six months after the Fall2023/Spring 2024 COVID-19 booster
  Evaluation of sustained cell mediated immunity against Covid-spike proteins. IFN-ϒ ELISpot, which detects both CD4 and CD8 T cell effectors, will be used to detect T-cell immunity to the Covid-spike protein or peptides.
Evaluate the persistence of memory B cell using memory B cell analysis. | during the Fall 2023 through Spring 2024 and at approximately six months after the Fall2023/Spring 2024 COVID-19 booster
  Evaluation of the persistence of memory B cell in approximately one-third of participants.
Sustained antibody concentration evaluating spike protein and receptor binding | during the Fall 2023 through Spring 2024 and at approximately six months after the Fall2023/Spring 2024 COVID-19 booster
  The NIH ELISA assay will be used to evaluate change in S and RBD (IgG and IgM) antibody titers.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ritter, MD, Principal Investigator — GI Alliance
Locations (4):
- United States (4):
  - Mayo Clinic Jacksonville, FL, Jacksonville, Florida
  - GI Alliance, Baton Rouge, Louisiana
  - GI Alliance, Southlake, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication.
Access Criteria: With researchers who provide a methodically sound proposal, to achieve aims in the approved proposal. Proposals should be directed to Tim.Ritter@GIAlliance.com.